CLINICAL TRIAL: NCT04233801
Title: A Phase III, Randomised, Double-blind, Placebo-controlled, Parallel Group Study of Empagliflozin (10 mg and 25 mg) Administered Orally Once Daily in Combination With Insulin With or Without up to Two Oral Anti-diabetic Agents for 24 Weeks in Chinese Type 2 Diabetic Patients With Insufficient Glycemic Control.
Brief Title: A Study to Test How Well Empagliflozin Works in Chinese Patients With Type 2 Diabetes Who Already Take Insulin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1245-0191
Record Dates: First submitted 2020-01-16; First posted 2020-01-18 (Actual); Results first posted 2023-12-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-03

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Empagliflozin 10 mg (Experimental): 1 table of 10 milligrams (mg) of Empagliflozin was administered orally once daily for a treatment period of 24 weeks.
  Before the first dose of randomised drug, all participants went through a 2-week open label placebo run-in period, taking Placebo tablets orally once daily.
  Interventions: Drug: Empagliflozin
- Empagliflozin 25 mg (Experimental): 1 table of 25 milligrams (mg) of Empagliflozin was administered orally once daily for a treatment period of 24 weeks.
  Before the first dose of randomised drug, all participants went through a 2-week open label placebo run-in period, taking Placebo tablets orally once daily.
  Interventions: Drug: Empagliflozin
- Placebo (Placebo Comparator): Matching placebo was administered orally once daily for a treatment period of 24 weeks.
  Before the first dose of randomised drug, all participants went through a 2-week open label placebo run-in period, taking Placebo tablets orally once daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Empagliflozin — Empagliflozin
  Arms: Empagliflozin 10 mg; Empagliflozin 25 mg
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a study in Chinese adults with type 2 diabetes. The study is open to people who take insulin but still have too high blood sugar levels. Participants may additionally be taking up to 2 other medicines for their diabetes. The purpose of this study is to find out whether empagliflozin taken together with insulin helps people with type 2 diabetes to better control their blood sugar.

The participants are in the study for about 7 months. During this time, they visit the study site about 8 times, 1 additional visit may be either a visit to the study site or a phone call. At the start of the study, participants are put into 3 groups by chance. Participants get either 10 mg empagliflozin tablets, or 25 mg empagliflozin tablets, or placebo tablets once a day. Placebo tablets look like empagliflozin tablets but do not contain any medicine.

The doctors regularly take blood samples from the participants. The changes in blood sugar levels are compared between the groups. The doctors also check the general health of the participants.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years and ≤75 years old at Visit 1;
* Chinese patient with diagnosis of Type 2 diabetes prior to Visit 1;
* A stable treatment with premixed Insulin (≥ 20IU/day) or basal insulin (≥ 16 IU/day) for at least 12 weeks prior to enrolment with or without up to two OADs

  * With maximum insulin dose of ≤ 1 unit/kg/day. Acceptable basal insulins should have duration of action up to 24 h such as insulin Degludec, insulin glargin, insulin detemir or NPH (neutral protamine hagedorn) insulin; Acceptable pre-mixed insulins could be once or twice daily posology only. The total insulin dose should not be changed by more than 20% of the baseline value within the 12 weeks prior to randomisation (Visit 3). Both human insulin & insulin analogue are acceptable;
  * If the patient is taking OADs, regimen has to be unchanged for at least 12 weeks prior to randomization (Visit 3);
  * If the patient is taking metformin, stable dose (at least 1500 mg daily or maximum tolerated dose) must be maintained for at least 12 weeks without dose adjustments prior to randomization (Visit 3);
* HbA1c ≥7.5% and ≤11.0% at Visit 1;
* Fasting C-peptide: >0.5 ng/mL (>166pmol/L) at Visit 1；
* 18.5 kg/m2 ≤ BMI ≤ 45 kg/m2 at Visit 1;
* Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial;
* Male or female patients. Women of childbearing potential (WOCBP) must be ready and able to use highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly. A list of contraception methods meeting these criteria is provided in the patient information.

Exclusion Criteria:

* Diagnosis of Type 1 diabetes;
* Patients receiving MDI insulin or insulin pump treatment;
* eGFR <45ml/min/1.73m2 calculated based on MDRD formula;
* Uncontrolled hyperglycemia [glucose level >13. 9 mmol/l after an overnight fast during placebo run-in];
* Severe hypoglycemia episode (event requiring the assistance of another person to actively administer carbohydrate, glucagon or other resuscitative actions) within 6 months prior to Visit 1;
* History of diabetic ketoacidosis or hyperosmolar non-ketotic coma. Myocardial infarction, stroke or transient ischaemic attack within 3 months prior to Visit 1;
* Bariatric surgery;
* Further criteria apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2022-03-03 (Actual); Study Completion 2022-03-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (24):
- China (24):
  - Peking University First Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - Beijing Pinggu Hospital, Beijing
  - The Second Hospital of Jilin University, Changchun
  - The third xiangya hospital of Central South University, Changsha
  - The First Hospital, Chongqing Medical University, Chongqing
  - Chongqing Three Gorges Central Hospital, Chongqing
  - Third Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - The Second Affiliated Hospital of Nanjing Medical University, Hangzhou
  - The Affiliated Hospital of Hangzhou Normal University, Hangzhou
  - Anhui Provincial Hospital, Hefei
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang
  - Jiangxi Provincial People's Hospital, Nanchang
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - The Second Affiliated Hospital to Nanchang University, Nanchang
  - The affiliated hospital of medicalcollege qingdao university, Qingdao
  - Tongren hospital, Shanghai Jiaotong University School of Medicine, Shanghai
  - Centre Hospital of Putuo District, Shanghai, Shanghai
  - Shanghai Fifth People's Hospital affiliated to Fudan University, Shanghai
  - Shengjing Hospital of China Medical University, Shenyang
  - Suzhou Municipal Hospital, Suzhou
  - The First Affiliated Hospital of Soochow University, Suzhou
  - Tianjin Medical University Chu Hisen-I Memorial Hospital, Tianjin

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and the primary manuscript is accepted for publishing, researchers can use this following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Also, Researchers can use the following link https://www.mystudywindow.com/msw/datasharing to find information in order to request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
  The data shared are the raw clinical study data sets
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by both the independent review panel and the sponsor, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a 'Data Sharing Agreement'.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was to determine the efficacy and safety of Empagliflozin added to insulin-treated type 2 diabetes patients.
Pre-assignment Details: 4 patients did not meet eligibility criteria but randomized and treated in this trial. The rest of the subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria.
Period: Overall Study
Arm/Group | Placebo | Empagliflozin 10 mg | Empagliflozin 25 mg
Started | 73 | 73 | 73
Completed | 73 | 71 | 69
Not Completed | 0 | 2 | 4
Not completed — Other than listed | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2 | 3

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The TS consisted of all patients who were randomised and treated with at least one dose of the study drug. The assignment of patients to treatment groups were based on the actual first study drug intake in the double-blind treatment period.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Empagliflozin 10 mg | Empagliflozin 25 mg | Total
Number analyzed (Participants) | 73 | 73 | 73 | 219
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.1 (8.0) | 59.9 (7.7) | 60.7 (9.1) | 60.2 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 30 | 33 | 100
  Male | 36 | 43 | 40 | 119
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 73 | 73 | 73 | 219
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Glycosylated haemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: Percentage of glycosylated hemoglobin] | 8.64 (0.81) | 8.64 (0.91) | 8.64 (0.88) | 8.64 (0.87)
Time since diagnosis of diabetes [Mean (Standard Deviation); unit: Years] | 14.14 (7.26) | 14.74 (7.01) | 15.05 (7.45) | 14.64 (7.22)
Background antidiabetic treatment [Count of Participants; unit: Participants]
  Insulin + Oral antidiabetic drug (OAD) | 60 | 59 | 59 | 178
  Insulin only | 13 | 14 | 14 | 41
Type of insulin [Count of Participants; unit: Participants]
  Basal | 32 | 38 | 34 | 104
  Pre-mixed | 41 | 35 | 39 | 115

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Haemoglobin A1c (HbA1c) at Week 24
Description: A restricted maximum likelihood (REML) based mixed model repeated measures (MMRM) approach was applied including treatment, background therapy, and visit as fixed classification effects, baseline HbA1c and baseline estimated glomerular filtration rate (eGFR) as the linear covariates, treatment by visit interaction, and baseline HbA1c by visit interaction.
Time Frame: At baseline (Week 0) and at Week 24
Population: Modified Intention-to-Treat (mITT) set: The mITT set consisted of all randomised patients who were treated with at least one dose of the study drug and had a baseline HbA1c assessment and at least one on-treatment glycosylated haemoglobin A1c (HbA1c) value. The assignment of patients to treatment groups were based on the planned randomised study drug at the time of randomisation.
Measure: Least Squares Mean (Standard Error); unit: Percentage of glycosylated hemoglobin
Arm/Group | Placebo | Empagliflozin 10 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 73 | 72 | 73
Percentage of glycosylated hemoglobin | -0.13 (0.10) | -1.12 (0.10) | -1.12 (0.10)
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 10 mg; Test type: Other — A restricted maximum likelihood (REML) based mixed model repeated measures (MMRM) approach was applied.The model included "baseline value for the corresponding endpoint" and its interaction with visit as additional covariates; p < 0.0001, Mixed model repeated measures; Adjusted mean = -0.99, 95% CI 2-sided [-1.28 to -0.71]
Statistical Analysis 2: Comparison: Placebo vs Empagliflozin 25 mg; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.0001, Mixed model repeated measures; Adjusted mean = -0.98, 95% CI 2-sided [-1.26 to -0.70]

2. Secondary Outcome: Percentage of Participants With HbA1c<7.0% at Week 24
Description: Percentage of participants with glycosylated haemoglobin A1c (HbA1c) <7.0% at Week 24 is reported.
Time Frame: At Week 24
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Empagliflozin 10 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 73 | 72 | 73
Percentage of participants | 8.2 | 16.7 | 30.1
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 10 mg; Test type: Other — Logistic regression including treatment, baseline Estimated glomerular filtration rate (eGFR), background therapy, and continuous baseline HbA1c; p = 0.1375, Regression, Logistic; Odds Ratio (OR) = 2.29, 95% CI 2-sided [0.77 to 6.83]
Statistical Analysis 2: Comparison: Placebo vs Empagliflozin 25 mg; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.0008, Regression, Logistic; Odds Ratio (OR) = 6.01, 95% CI 2-sided [2.11 to 17.10]

3. Secondary Outcome: Change in Body Weight From Baseline to Week 24
Description: Change in body weight from baseline to Week 24 is reported. A restricted maximum likelihood (REML) based mixed model repeated measures (MMRM) approach was applied including baseline body weight, and its interaction with visit.
Time Frame: At baseline (Week 0) and at Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Kilogram
Arm/Group | Placebo | Empagliflozin 10 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 73 | 72 | 73
Kilogram | 0.01 (0.23) | -1.99 (0.24) | -1.31 (0.24)
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 10 mg; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.0001, Mixed model repeated measures; Adjusted mean = -2.00, 95% CI 2-sided [-2.66 to -1.34]
Statistical Analysis 2: Comparison: Placebo vs Empagliflozin 25 mg; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.0001, Mixed model repeated measures; Adjusted mean = -1.32, 95% CI 2-sided [-1.96 to -0.67]

4. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) at Week 24
Description: A restricted maximum likelihood (REML) based mixed model repeated measures (MMRM) approach was applied including baseline SBP and its interaction with visit.
Time Frame: At baseline (Week 0) and at Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Millimetre of mercury (mmHg)
Arm/Group | Placebo | Empagliflozin 10 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 73 | 72 | 73
Millimetre of mercury (mmHg) | -1.95 (1.38) | -5.56 (1.49) | -2.96 (1.46)
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 10 mg; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0774, Mixed model repeated measures; Adjusted mean = -3.60, 95% CI 2-sided [-7.61 to 0.40]
Statistical Analysis 2: Comparison: Placebo vs Empagliflozin 25 mg; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.6160, Mixed model repeated measures; Adjusted mean = -1.01, 95% CI 2-sided [-4.98 to 2.96]

5. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure (DBP) at Week 24
Description: A restricted maximum likelihood (REML) based mixed model repeated measures (MMRM) approach was applied including baseline DBP and its interaction with visit.
Time Frame: At baseline (Week 0) and at Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Millimetre of mercury (mmHg)
Arm/Group | Placebo | Empagliflozin 10 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 73 | 72 | 73
Millimetre of mercury (mmHg) | -1.59 (0.78) | -3.37 (0.84) | -0.94 (0.83)
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 10 mg; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.1222, Mixed model repeated measures; Adjusted mean = -1.78, 95% CI 2-sided [-4.05 to 0.48]
Statistical Analysis 2: Comparison: Placebo vs Empagliflozin 25 mg; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.5687, Mixed model repeated measures; Adjusted mean = 0.65, 95% CI 2-sided [-1.59 to 2.89]

6. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 24
Description: A restricted maximum likelihood (REML) based mixed model repeated measures (MMRM) approach was applied including baseline FPG and its interaction with visit.
Time Frame: At baseline (Week 0) and at Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Milligrams per deciliter (mg/dL)
Arm/Group | Placebo | Empagliflozin 10 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 73 | 72 | 73
Milligrams per deciliter (mg/dL) | -5.56 (3.67) | -25.61 (3.97) | -29.69 (3.90)
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 10 mg; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0003, Mixed model repeated measures; Adjusted mean = -20.05, 95% CI 2-sided [-30.73 to -9.38]
Statistical Analysis 2: Comparison: Placebo vs Empagliflozin 25 mg; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.0001, Mixed model repeated measures; Adjusted mean = -24.13, 95% CI 2-sided [-34.72 to -13.54]

7. Secondary Outcome: Change From Baseline in 2-hour Post-prandial Glucose (PPG) at Week 24
Description: The Analysis of covariance (ANCOVA) model included treatment and background therapy as classification effects, baseline PPG and baseline Estimated glomerular filtration rate (eGFR) as the linear covariates.
Time Frame: At baseline (Week 0) and at Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Milligrams per deciliter (mg/dL)
Arm/Group | Placebo | Empagliflozin 10 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 73 | 72 | 73
Milligrams per deciliter (mg/dL) | 3.27 (7.53) | -53.05 (8.14) | -57.44 (7.89)
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 10 mg; Test type: Other — The Analysis of covariance (ANCOVA) model included treatment and background therapy as classification effects, baseline PPG and baseline Estimated glomerular filtration rate (eGFR) as the linear covariates; p < 0.0001, ANCOVA; Adjusted mean = -56.32, 95% CI 2-sided [-78.22 to -34.41]
Statistical Analysis 2: Comparison: Placebo vs Empagliflozin 25 mg; Test type: Other — [test comment as in outcome 7, analysis 1]; p < 0.0001, ANCOVA; Adjusted mean = -60.71, 95% CI 2-sided [-82.31 to -39.11]

8. Secondary Outcome: Number of Participants With Confirmed Hypoglycaemic Events
Description: Confirmed hypoglycemic events refer to the hypoglycaemic events with a plasma glucose value of ≤70 milligrams per deciliter (mg/dL) or where assistance was required.
Time Frame: From first administration of the initial randomised study medication to last intake of study medication + 7 days (inclusive), up to 176 days.
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Empagliflozin 10 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 73 | 73 | 73
Participants | 8 | 13 | 7
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 10 mg; Test type: Other; p = 0.2422, Regression, Logistic; Logistic regression including treatment and continuous baseline glycosylated haemoglobin A1c (HbA1c); Odds Ratio (OR) = 1.76, 95% CI 2-sided [0.68 to 4.55] — Odds ratio used Placebo as the reference group
Statistical Analysis 2: Comparison: Placebo vs Empagliflozin 25 mg; Test type: Other; p = 0.7661, Regression, Logistic; Logistic regression including treatment and continuous baseline glycosylated haemoglobin A1c (HbA1c); Odds Ratio (OR) = 0.85, 95% CI 2-sided [0.29 to 2.50] — Odds ratio used Placebo as the reference group

9. Secondary Outcome: Number of Participants With Adjudicated Diabetic Ketoacidosis (DKA) Events
Description: The risk of DKA had to be considered in the event of non-specific symptoms such as nausea, vomiting, anorexia, abdominal pain, excessive thirst, difficulty in breathing, confusion, unusual fatigue or sleepiness. In case of a suspected DKA, the investigator was to ensure that appropriate tests were performed at the earliest opportunity according to 2017 China Type 2 diabetes mellitus (T2DM) guidelines.
  An independent external Clinical event committee (CEC) was established to adjudicate centrally and in a blinded fashion events suspected of DKA and certain hepatic events.
  DKA was investigated using both broad and narrow Boehringer Ingelheim customised MedDRA query (BIcMQs).
Time Frame: as for outcome 8
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Empagliflozin 10 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 73 | 73 | 73
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: For Run-in period group: from first dose of open label placebo till end of run-in period, up to 2 weeks. For the other groups: From first administration of the initial randomised study medication to last intake of study medication + 7 days (inclusive), up to 176 days.
Description: Treated set (TS): The TS consisted of all patients who were randomised and treated with at least one dose of the study drug. The assignment of patients to treatment groups were based on the actual first study drug intake in the double-blind treatment period.
Groups:
- Run-in Period: Before the first dose of randomised drug, all participants went through a 2-week open label placebo run-in period, taking Placebo tablet orally once daily.
  This group includes all participants who participated the run-in period.
Arm/Group | Placebo | Empagliflozin 10 mg | Empagliflozin 25 mg | Run-in Period
All-Cause Mortality (participants affected / at risk) | 0/73 | 0/73 | 0/73 | 0/219
Serious Adverse Events (participants affected / at risk) | 6/73 | 10/73 | 7/73 | 2/219
Other Adverse Events (participants affected / at risk) | 39/73 | 27/73 | 27/73 | 46/219
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=73) | Empagliflozin 10 mg (N=73) | Empagliflozin 25 mg (N=73) | Run-in Period (N=219)
Angina unstable (Cardiac disorders) | 0 | 0 | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 1 | 1 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Hyperparathyroidism (Endocrine disorders) | 0 | 1 | 0 | 0
Thyroid mass (Endocrine disorders) | 0 | 1 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 1 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Appendicitis perforated (Infections and infestations) | 0 | 0 | 1 | 0
Complicated appendicitis (Infections and infestations) | 0 | 0 | 1 | 0
Erysipelas (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0
Meningitis viral (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Benign anorectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1 | 0
Parkinson's disease (Nervous system disorders) | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=73) | Empagliflozin 10 mg (N=73) | Empagliflozin 25 mg (N=73) | Run-in Period (N=219)
Upper respiratory tract infection (Infections and infestations) | 5 | 4 | 4 | 3
Urinary tract infection (Infections and infestations) | 10 | 6 | 6 | 10
Electrocardiogram T wave abnormal (Investigations) | 5 | 1 | 2 | 0
Protein urine present (Investigations) | 4 | 2 | 3 | 15
Hyperglycaemia (Metabolism and nutrition disorders) | 7 | 0 | 3 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 | 4 | 4 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 11 | 15 | 11 | 9
Diabetic nephropathy (Renal and urinary disorders) | 6 | 0 | 1 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results.

Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days.

BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-04-20): https://cdn.clinicaltrials.gov/large-docs/01/NCT04233801/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-12): https://cdn.clinicaltrials.gov/large-docs/01/NCT04233801/SAP_001.pdf